CLINICAL TRIAL: NCT05984329
Title: Tonic Versus Burst DR(TM) Epidural Motor Cortex Stimulation for Neuropathic Pain : a Double-blind, Crossover, Comparative Study
Brief Title: Tonic Versus Burst DR(TM) Epidural Motor Cortex Stimulation for Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN872022/CHUSTE
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-07

CONDITIONS: Neuropathic Pain
Keywords: Motor cortex stimulation; neuropathic pain; Burst DR(TM) waveform
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tonic then Burst DR(TM): Tonic Motor Cortex Stimulation (MCS) for 3 months then Burst DR(TM) MCS for 3 months
  Interventions: Other: Retrospective analysis of patients' choice
- Burst DR(TM) then tonic: Burst DR(TM) MCS for 3 months then tonic MCS for 3 months
  Interventions: Other: Retrospective analysis of patients' choice

INTERVENTIONS:
Other: Retrospective analysis of patients' choice — Retrospective analysis of patients' choice of tonic or Burst DR(TM) waves for their analgesic effect.

SUMMARY:
Epidural stimulation of the primary motor cortex (PMC) is indicated for the relief of neuropathic pain refractory to pharmacological treatment.

DETAILED DESCRIPTION:
The main objective of this study is to compare the analgesic effect of two distinct waveforms (i.e. tonic versus Burst DR(TM)) delivered by an epidural stimulator of the (primary) motor cortex in patients suffering from neuropathic pain resistant to the best pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from neuropathic pain refractory to best pharmacological treatment, operated on for MCS with an internal pulse generator (IPG) capable of delivering both tonic and Burst DR(TM) stimulation waveforms.

Exclusion Criteria:

* Patients under 18 years old ; pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MCS patients.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Percentage of pain relief | 6 months
  Percentage of analgesic relief compared with baseline (i.e. preoperative pain level)

SECONDARY OUTCOMES:
Antalgic drugs intake | 6 months
  Modification of pharmacological treatment doses (analgesics)

CONTACTS AND LOCATIONS:
Overall Officials: François VASSAL, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No